CLINICAL TRIAL: NCT00872547
Title: Prospective, International Multi-centre, Uncontrolled, Post Marketing Surveillance Study to Monitor the Long-term Performance of a Large Metal-on-Metal (MoM) Bearing Comprising a DePuy ASR™ Cup in Conjunction With Either a DePuy ASR™ Hip Resurfacing Femoral Component or a DePuy ASR™ XL Head in Subjects With Indications Suitable for Either a Primary Resurfacing Arthroplasty or Primary Total Hip Arthroplasty
Brief Title: Multi-Centre Study to Assess the Long-term Performance of the DePuy ASR™ System in Resurfacing and Primary Total Hip Replacement
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: DePuy discontinued this product in 4Q2009. At the time of this decision DePuy reviewed all clinical studies for this product and decided to close this Study
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT05/18
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-07

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Post-traumatic Arthritis; Collagen Disorders; Avascular Necrosis; Nonunion of Femoral Fractures; Congenital Hip Dysplasia; Slipped Capital Femoral Epiphysis
Keywords: Hip; Resurfacing; Metal-on-Metal; Large Heads; XL Head; ASR - osteoarthritis (primary)
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Collagen Diseases; Osteonecrosis; Hip Dislocation, Congenital; Slipped Capital Femoral Epiphyses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Resurfacing system
  Interventions: Device: DePuy ASR™ Hip System
- 2 (Active Comparator): Large Metal-on-Metal Total Hip Replacement
  Interventions: Device: DePuy ASR™ XL Head / ASR™ Acetabular Cup System

INTERVENTIONS:
Device: DePuy ASR™ Hip System — Resurfacing system
  Arms: 1
Device: DePuy ASR™ XL Head / ASR™ Acetabular Cup System — Large Metal-on-Metal Total Hip Replacement
  Arms: 2

SUMMARY:
The purpose of this study is to monitor the performance of a large metal-on-metal bearing from the DePuy ASR™ System in the treatment of patients with hip joint disease requiring hip resurfacing surgery or a total hip replacement. Patients who enter the study will be evaluated at regular intervals following hip surgery using patient, clinical and x-ray assessments.

The Study was terminated with effect from 30th November 2011 following the completion of 2 year follow up assessments for those patients remaining in the study.

Please note that prior to this decision DePuy voluntarily recalled the ASR products on 24 August 2010. Additional information regarding this voluntary recall and the follow-up of patients affected by the recall can be found at the following links http://www.mhra.gov.uk/Publications/Safetywarnings/MedicalDeviceAlerts/CON155761 and http://www.depuy.com/countries_list.

ELIGIBILITY:
General Inclusion Criteria:

i) Male or female subjects, aged between 18 and 65 years inclusive.

ii) Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.

iii) Subjects, who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.

Inclusion Criteria for DePuy ASR™ Resurfacing system:

i) Subjects with primary osteoarthritis indicated for standard MoM hip resurfacing arthroplasty with cementless fixation in the acetabulum.

Inclusion Criteria for ASR™ XL Head system:

i) Subjects whose bone morphology and bone quality mean that standard MoM hip resurfacing arthroplasty is not indicated, but for whom cementless fixation in the acetabulum and receipt of a large MoM bearing are still possible.

General Exclusion Criteria:

i) Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.

ii) Subjects with compromised renal function defined as those whose measured values lie outside the normal range for a particular investigational site.

iii) Subjects with proven metal sensitivity.

iv) Subjects with infectious, highly communicable diseases, which may limit follow-up i.e. Active tuberculosis, hepatitis, immuno-compromised conditions, etc.

v) Women who are pregnant or who intend to become pregnant within 2 years of surgery.

vi) Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.

vii) Subjects who have participated in a clinical study with an investigational product in the last 6 month(s).

viii) Subjects who are currently, or have been in the last 12 months, participating in a clinical study which involves exposure to ionising radiation.

ix) Subjects who are currently involved in any injury litigation claims.

x) Subjects who are undergoing corticosteroid treatment.

xi) Subjects with active or recent joint sepsis.

Additional Exclusion Criteria for DePuy ASR™:

i) Subjects with proven significant osteoporosis and poor bone quality.

ii) Subjects with marked atrophy or deformity in the upper femur, skeletal immaturity, or where loss of musculature or neuromuscular disease would render the procedure unjustifiable.

iii) Subjects whose anatomical CCD angle is below 120°.

iv) Subjects who have undergone irradiation of the affected hip.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2006-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Kaplan-Meier survivorship calculated at the five-year time-point | 5yrs

SECONDARY OUTCOMES:
Annual Kaplan-Meier survivorship calculations | Annually
Harris Hip Score | 3mths, 1yr, 2yrs, 5yrs, 10yrs, and 15yrs post-surgery
Radiographic analysis | 3mths, 1yr, 2yrs, 5yrs, 10yrs, and 15yrs post-surgery
Oxford Hip Score | 3mths, 6mths and annually post-surgery
UCLA Activity Score | 3mths, 6mths and annually post-surgery
Hip Outcome Score | 3mths, 6mths and annually post-surgery
EuroQol EQ-5D | 3mths, 6mths and annually post-surgery

CONTACTS AND LOCATIONS:
Locations (8):
- University Clinic for Orthopaedics and Orthopaedic Surgery - LKH, Graz, Austria
- Znojmo Hospital, Znojmo, Czechia
- Coxa, Hospital for Joint Replacement, Tampere, Finland
- Klinikum der Universität zu, Cologne, Germany
- Elverum Hospital, Elverum, Norway
- Hospital Curry Cabral, Lisbon, Curry Cabral, Portugal
- Kant. Spital Sursee-Wolhusen, Wolhusen, Switzerland
- Royal Berkshire Hospital, UK, Reading, Berkshire, United Kingdom